CLINICAL TRIAL: NCT02239120
Title: Randomized, Double-blind, Evaluation in Secondary Stroke Prevention Comparing the EfficaCy and Safety of the Oral Thrombin Inhibitor Dabigatran Etexilate (110 mg or 150 mg, Oral b.i.d.) Versus Acetylsalicylic Acid (100 mg Oral q.d.) in Patients With Embolic Stroke of Undetermined Source (RESPECT ESUS)
Brief Title: Dabigatran Etexilate for Secondary Stroke Prevention in Patients With Embolic Stroke of Undetermined Source (RE-SPECT ESUS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 1160.189; 2013-003444-24 (EudraCT Number)
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Stroke; Secondary Prevention
MeSH Terms: conditions — Stroke | interventions — Dabigatran

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- dabigatran etexilate 110 or 150 mg (Experimental): Patients will be assigned Dabigatran 150 mg b.i.d. (unless they are 75 years or older, or have a Creatinine Clearance (CrCl) of greater than or equal to 30 to less than 50ml/min (or experience GI bleed during trial), in which case they will receive Dabigatran 110 mg b.i.d.). All patients in this arm will also receive ASA placebo (q.d.)
  Interventions: Drug: optional ASA as comedication; Drug: placebo to ASA; Drug: dabigatran etexilate
- ASA 100 mg (Active Comparator): All patients will receive blinded ASA 100 mg q.d. and dabigatran placebo 150 mg b.i.d. (unless they are 75 years or older, or have a CrCl of greater than or equal to 30 to less than 50ml/min (or experience GI bleed during trial), in which case they will receive placebo Dabigatran 110 mg b.i.d
  Interventions: Drug: placebo to optional ASA as comedication; Drug: placebo to dabigatran etexilate; Drug: ASA 100 mg

INTERVENTIONS:
Drug: optional ASA as comedication — optional concomitant treatment which can be used for patients with coronary artery disease. It is not required for these pts.
  Arms: dabigatran etexilate 110 or 150 mg
Drug: placebo to ASA — placebo to comparator drug
  Arms: dabigatran etexilate 110 or 150 mg
Drug: placebo to optional ASA as comedication — optional concomitant treatment which can be used for patients with coronary artery disease. It is not required for these pts.
  Arms: ASA 100 mg
Drug: placebo to dabigatran etexilate — placebo
  Arms: ASA 100 mg
Drug: ASA 100 mg — active comparator drug
  Arms: ASA 100 mg
Drug: dabigatran etexilate — active drug
  Arms: dabigatran etexilate 110 or 150 mg

SUMMARY:
This trial will enroll approximately 6,000 patients with recent embolic stroke of unknown source (ESUS). Patients will be randomized to dabigatran or acetylsalicyclic acid (ASA) (1:1 ratio) and have visits every three months. The study doctor may prescribe blinded concomitant ASA for pts with coronary artery disease but this is not mandatory. All Adverse Events (AEs), Serious Adverse Events (SAEs), outcome events will be recorded. The trial will conclude when the required number of stroke events are positively adjudicated which is estimated to take 3 years (including 2.5 years of enrollment).

ELIGIBILITY:
Inclusion criteria:

* Ischemic stroke with a brain lesion visualized by neuroimaging (either brain Computed Tomography (CT) or Magnetic Resonance Image (MRI)). The visualized stroke is a non-lacunar infarct , e.g. involving the cortex or >1.5 cm (>2.0 cm if measured on MRI diffusion-weighted images) in largest diameter if exclusively subcortical.Visualization by CT usually requires delayed imaging >24-48 hours after stroke onset.
* The index stroke must have occurred either up to 3 months before randomization (Modified Rankin Scale(mRS) <=3 at randomization) or up to 6 months before randomization (mRS <=3 at randomization) in selected patients that are >= 60 years plus at least one additional risk factor for recurrent stroke.
* Arterial imaging or cervical plus Transcranial Doppler (TCD) ultrasonography does not show extra-cranial or intracranial atherosclerosis with >= 50% luminal stenosis in artery supplying the area of acute ischemia.
* As evidenced by cardiac monitoring for >= 20 hours with automated rhythm detection, there is absence of AF > 6 minutes in duration (within a 20 hour period, either as single episode or cumulative time of multiple episodes).

Further inclusion criteria apply.

Exclusion criteria:

* Modified Rankin Scale of >=4 at time of randomization or inability to swallow medications.
* Major risk cardioembolic source of embolism such as: a) intracardiac thrombus as evidenced by transthoracic or transesophageal echocardiography, b) paroxysmal, persistent or permanent Atrial fibrillation (AF), c) atrial flutter, d) prosthetic cardiac valve (mitral or aortic, bioprosthetic or mechanical), e) atrial myxoma, f) other cardiac tumors, g) moderate or severe mitral stenosis, h) recent (< 4weeks) myocardial infarction, i) valvular vegetations, or j) infective endocarditis.
* Any indication that requires treatment with an anticoagulant as per Investigator's judgment.
* History of atrial fibrillation (unless it was due to reversible causes such as hyperthyroidism or binge drinking, and has been permanently resolved).
* Other specific stroke etiology (i.e. cerebral arteritis or arterial dissection, migraine with aura/vasospasm, drug abuse).
* Renal impairment with estimated creatinine clearance (as calculated by Cockcroft-Gault equation) <30mL/min at screening, or where Investigator expects creatinine clearance is likely to drop below 30mL/min during the course of the study.

Further exclusion criteria apply.

Ages: 18 Years to 150 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5390 (Actual)
Dates: Start 2014-11-27 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (566):
- United States (110):
  - Bronislava Shafran, MD PC, Phoenix, Arizona
  - Westside Medical Associates of Los Angeles, Beverly Hills, California
  - TriWest Research Associates, LLC, El Cajon, California
  - University of California, Fresno, California
  - Glendale Adventist Medical Center, Glendale, California
  - Collaborative Neuroscience Network, LLC (CNS), Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Huntington Hospital, Pasadena, California
  - University of California, San Diego, California
  - University of California, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Colorado Neurological Institute, Englewood, Colorado
  - University of Colorado Denver, Fort Collins, Colorado
  - St. Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Tenet Florida Physician Services, Boynton Beach, Florida
  - Nova Clinical Research, LLC, Bradenton, Florida
  - Broward Health North, Deerfield Beach, Florida
  - Center for Advanced Research Excellence, Hialeah, Florida
  - Bruce W. Carter, Miami VA Healthcare System, Miami, Florida
  - University of Miami, Miami, Florida
  - Bay Neurological Institute, Panama City, Florida
  - Carol L Pappas, MD PhD PA, St. Petersburg, Florida
  - University of South Florida, Tampa, Florida
  - Vero Beach Neurology and Research Institute, Vero Beach, Florida
  - Palm Beach Neuroscience Institute, West Palm Beach, Florida
  - Augusta University, Augusta, Georgia
  - WellStar Medical Group - Neurosurgery, Marietta, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Medical Center-Neurology, Boise, Idaho
  - Northwest Heart Clinical Research, LLC, Arlington Heights, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Medicoricium, LLC, Fairview Heights, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Quincy Physicians and Surgeons Clinic, S.C., Quincy, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Community Clinical Research Center, Anderson, Indiana
  - Ruan Neurology Clinic and Research Center, Des Moines, Iowa
  - Associates in Neurology, PSC, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Alexandria Cardiology Clinic, Alexandria, Louisiana
  - Culicchia Neurological Clinic, Marrero, Louisiana
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - McLaren Flint, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health Medical Center, Grand Rapids, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - The Duluth Clinic dba Essentia Health Duluth Clinic, Duluth, Minnesota
  - Abbott Northwestern Hospital, Radiology Department, Minneapolis, Minnesota
  - HealthPartners Neuroscience Center, Saint Paul, Minnesota
  - Jackson Heart Clinic, P.A., Jackson, Mississippi
  - Boone Hospital Center, Columbia, Missouri
  - University of Missouri Health System, Columbia, Missouri
  - SSM Health St. Clare Hospital, Fenton, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - St. Louis Heart and Vascular, P.C., St Louis, Missouri
  - The Nebraska Medical Center, Omaha, Nebraska
  - Renown Institute for Neurosciences, Reno, Nevada
  - NYC Health + Hospitals/Coney Island, Brooklyn, New York
  - New York Presbyterian Hudson Valley Hospital, Cortlandt Manor, New York
  - UHS Wilson Medical Center,Office of Clin Trials, Johnson City, New York
  - North Shore University Hospital, Manhasset, New York
  - Winthrop University Hospital, Mineola, New York
  - Mount Sinai Beth Israel, New York, New York
  - Novant Health Neurology Specialists, Charlotte, North Carolina
  - Duke Clinic 1L, Durham, North Carolina
  - Cone Health System, Greensboro, North Carolina
  - Novant Health Neurology Hickory, Hickory, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Altru Health System, Grand Forks, North Dakota
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Holzer Clinic LLC, Gallipolis, Ohio
  - Advanced Neurology Associates, Youngstown, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - Veterans Affairs Portland Health Care System, Portland, Oregon
  - Sacred Heart Medical Center at RiverBend, Springfield, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Methodist University Hospital, Memphis, Tennessee
  - Centennial Heart Cardiovascular Consultants, LLC, Nashville, Tennessee
  - Saint Thomas Health, Nashville, Tennessee
  - Seton Medical Center Austin, Austin, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Bhupesh Dihenia, M.D.,P.A., Lubbock, Texas
  - University of Vermont, Burlington, Vermont
  - Virginia Commonwealth University, Richmond, Virginia
  - Carilion Riverside, Roanoke, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Neuroscience Institute, Seattle, Washington
  - Marshall University, Huntington, West Virginia
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin, Madison, Wisconsin
- Argentina (6):
  - STAT Research, CABA
  - Fundación Favaloro, CABA
  - Hospital Italiano de Buenos Aires, CABA
  - Clinica Coronel Suarez SA, Coronel Suárez
  - Instituto Médico DAMIC S.R.L., Córdoba
  - Hospital Privado de Comunidad, Mar del Plata
- Australia (13):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Kanwal Medical Complex, Kanwal, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Calvary North Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Austin Health, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Alfred Health, Victoria, Victoria
- Austria (7):
  - LKH-Univ. Hospital Graz, Graz
  - Medical University of Innsbruck, Innsbruck
  - Kepler Univ. Klinikum Linz, Linz
  - KH d. Barmherzigen Brüder Linz, Neurologie, Linz
  - Universitätsklinikum Tulln, Abteilung für Neurologie, Tulln
  - Hosp.Hietzing with Neuro.Centr Rosenhuegel,II Neuro.dep,Wien, Vienna
  - Wilhelminenspital, Vienna
- Belgium (15):
  - Aalst - HOSP Onze-Lieve-Vrouw, Aalst
  - Arlon - HOSP Sud Luxembourg - Vivalia, Arlon
  - AZ Sint-Jan Brugge, Bruges
  - Brussels-UNIV Brugmann -Horta, Brussels
  - Brussels - HOSP Europe (Ste-Elisabeth), Brussels
  - Brussels - UNIV Saint-Luc, Brussels
  - UNIV UZ Gent, Ghent
  - Kortrijk - HOSP AZ Groeninge Kennedylaan, Kortrijk
  - UZ Leuven, Leuven
  - Liège - HOSP St-Joseph, Liège
  - Roeselare - HOSP AZ Delta, Roeselare
  - Rumst - HOSP AZ Heilige Familie, Rumst
  - Sint-Truiden - HOSP St-Trudo (St-Jozef), Sint-Truiden
  - Wilrijk - HOSP GZA (St-Augustinus), Wilrijk
  - Yvoir - UNIV UCL de Mont-Godinne, Yvoir
- Brazil (6):
  - Hospital Clinicas de Botucatu, Botucatu
  - Instituto de Medicina Flumignano, Curitiba
  - Clinica Neurologica e Neurocirurgica de Joinvile, Joinvile
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - H.C.da Fac. de Medicina de Ribeirao Preto, Ribeirão Preto
  - Hospital Quinta D¿Or, Rio de Janeiro
- Canada (17):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital (University of Alberta), Edmonton, Alberta
  - Grey Nuns Hospital, Edmonton, Alberta
  - Prairie Mountain Health, Brandon, Manitoba
  - Hopital Notre-Dame du CHUM, Montreal, Migration Data
  - Jewish General Hospital, Montreal, Migration Data
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Eastern Health (MUN), St. John's, Newfoundland and Labrador
  - Victoria Hospital (LHSC), London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - CSSS de Chicoutimi, Chicoutimi, Quebec
  - Hopital Charles - LeMoyne, Greenfield Park, Quebec
  - Montreal General Hospital - McGill University Health Centre, Montreal, Quebec
  - St Jerome Medical Research Inc., Saint-Jérôme, Quebec
  - CHUS Fleurimont, Sherbrooke, Quebec
  - CHU de Quebec-Universite Laval Research Centre, Québec
- Chile (3):
  - Clínica Alemana de Santiago S.A., Santiago
  - Clínica Dávila, Santiago
  - Clinica Alemana de Temuco, Temuco
- China (22):
  - Beijing Tiantan Hospital affiliated to Cap Med University, Beijing
  - Peking University Third Hospital, Beijing
  - First Hospital of Jilin University, Changchun
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - First Affiliated Hospital of Guangzhou University of TCM, Guangzhou
  - The First Affiliated Hospital of Jinan University, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - 2nd Affiliated Hosp Zhejiang University College of Medical, Hangzhou
  - Zhejiang Hospital, Hangzhou
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou
  - Zhejiang University School of Medicine SIR RUN RUN SHAW Hospital, Hangzhou
  - Jinlin Central Hospital, Jilin
  - The Second Affiliated Hospital to Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - QingDao Municipal Hospital, Qingdao
  - The affiliated hospital of medicalcollege qingdao university, Qingdao
  - Huashan Hospital, Fudan University, Shanghai
  - Tongji Hospital, Tongji University, Shanghai
  - General Hospital of Shenyang Military Region, Shenyang
  - First Affiliated Hospital of Xiamen University, Xiamen
  - Affiliated Hospital, Xuzhou Medical college, Xuzhou
- Colombia (4):
  - Servicios Médicos Muñoz Solano, Bogotá
  - Sociedad de Cirugia de Bogota Hospital de San José, Bogotá
  - Fundación Valle del Lili, Cali
  - Fundación Cardiovascular de Colombia, Floridablanca
- Croatia (4):
  - General Hospital Varazdin, Varaždin
  - Clin.Hosp.Centre Zagreb,Cerebrovascul.disease w/ intens.care, Zagreb
  - University hospital center Zagreb, Zagreb
  - Univ. Hosp. Sisters of Mercy, Neurology Clinic, Zagreb, Zagreb
- Czechia (6):
  - Cerebrovascular site, private prac., Brno, Brno
  - Hospital Jihlava, Jihlava
  - University Hospital Olomouc, Olomouc
  - Cerebrovascular site, Ostrava, Ostrava
  - University Hospital Motol, Prague
  - Hospital Homolka, Prague, Prague
- Estonia (4):
  - East Estonia Central Hospital, Neurology Dept, Ahtme, Ahtme
  - West Tallinn Central Hospital, Neurology Dept., Tallinn
  - North Estonia Medical Centre Foundation, Tallin, Tallinn
  - Tartu University Hospital, Tartu
- France (13):
  - HOP Pays d'Aix, Aix-en-Provence
  - HOP de Bayonne, Bayonne
  - HOP Jean Minjoz, Besançon
  - HOP Pellegrin, Bordeaux
  - HOP de la Cavale Blanche, Brest
  - HOP Pierre Wertheimer, Bron
  - HOP Côte de Nacre, Caen
  - HOP Grenoble, Neuro, Grenoble, Grenoble
  - HOP Roger Salengro, Lille
  - HOP Mercy, Metz
  - HOP Paris Saint-Joseph, Paris
  - GHU Paris Psychiatrie et Neurosciences, Paris
  - HOP Purpan, Toulouse
- Germany (69):
  - Klinikum Altenburger Land GmbH, Altenburg
  - Neurologische Klinik GmbH, Bad Neustadt, Bad Neustadt an der Saale
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Evangelisches Klinikum Bethel gGmbH, Bielefeld
  - Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil gGmbH, Bochum
  - St. Josef- und St. Elisabeth-Hospital gGmbH, Bochum
  - Gesundheit Nord gGmbH | Klinikverbund Bremen, Bremen
  - Klinikum Bremerhaven, Bremen
  - Krankenhäuser Buchholz und Winsen gGmbH, Buchholz
  - Allgemeines Krankenhaus, Celle, Celle
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Klinikum Coburg gGmbH, Coburg
  - Universitätsklinikum Köln (AöR), Cologne
  - Klinikzentrum Mitte, Dortmund, Dortmund
  - Städtisches Klinikum Dresden, Dresden
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Marien-Hospital, Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Alfried Krupp Krankenhaus Essen, Essen
  - Universitätsklinikum Essen AöR, Essen
  - Klinikum Frankfurt Höchst GmbH, Frankfurt
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Klinikum Friedrichshafen, Friedrichshafen
  - Klinikum Fulda gAG, Fulda
  - Evangelische Klinik Gelsenkirchen, Gelsenkirchen
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - Universitätsmedizin Greifswald, Greifswald
  - Bezirkskrankenhaus, Günzburg, Günzburg
  - Asklepios Klinik St. Georg, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Harburg, Hamburg
  - Asklepios Klinik Wandsbek, Hamburg
  - Asklepios Klinik Barmbek, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Klinikum Hanau GmbH, Hanau
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Klinikum Idar-Oberstein, Idar-Oberstein
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - Universitätsklinikum Magdeburg AöR, Magdeburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Gießen und Marburg GmbH, Marburg
  - Elblandklinikum Meißen, Meißen
  - Johannes Wesling Klinikum, Minden
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Ökumenisches Hainich Klinikum gGmbH, Mühlhausen
  - Klinikum der Universität München - Campus Großhadern, München
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Universitätsklinikum Münster, Münster
  - Klinikum Nürnberg, Nuremberg
  - Sana Klinikum Offenbach GmbH, Offenbach
  - Klinikum Osnabrück GmbH, Osnabrück
  - Universitätsklinikum Regensburg, Regensburg
  - Nordwest-Krankenhaus Sanderbusch gGmbH, Sande
  - Kreisklinikum Siegen GmbH, Siegen
  - Bürgerhospital, Stuttgart, Stuttgart
  - Nervenklinik Teupitz, Teupitz, Teupitz
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Universitätsklinikum Tübingen, Tübingen
  - RKU - Universitäts- und Rehabilitationskliniken Ulm gGmbH, Ulm
  - Sophien- und Hufeland-Klinikum gGmbH, Weimar
  - Helios Dr. Horst Schmidt Kliniken Wiesbaden, Wiesbaden
  - Universitätsklinikum Würzburg, Würzburg
- Greece (7):
  - Univ.Hosp. of Alexandroupolis, Alexandroupoli
  - Gen.Hosp.of Ath.Evangelismos, Athens
  - Attikon University Hospital, Athens
  - Gen.Univ. Hosp. of Herakleion, Heraklion
  - General University Hospital of Larissa, Larissa
  - Univ. Gen. Hosp. of Patras, Pátrai
  - Univ.Gen.Hosp. of Thessaloniki, Thessaloniki
- Hong Kong (3):
  - Prince of Wales Hospital, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Hungary (6):
  - Semmelweis University, Budapest
  - National Instit.of Neurosciences,Neurology Dept,Budapest, Budapest
  - Univ. Debrecen Medical Health Science Center, Neurology Dept, Debrecen
  - Pest Megyei Flor Ferenc Hospital, Kistarcsa
  - CRU Hungary Ltd, Private Practice, Miskolc, Miskolc
  - Univ. of Pecs Clinic for Neurology, Pécs
- India (11):
  - St. Johns medical College and Hospital, Bangalore
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - Lalitha Super Specialities Hospital, Guntur
  - Nizam's Institute of Medical Sciences, Hyderabad
  - Shree Krishna Hospital and Research Centre, Karamsad
  - Caritas Hospital, Kottayam
  - Mangala Hospital and Mangala Kidney Foundation, Mangalore
  - LTMMC & GH Medical College,, Mumbai
  - Magnum Heart Institute, Nashik
  - All India Institute of Medical Sciences, New Delhi
  - Sahyadri Speciality Hospital, Pune
- Israel (4):
  - Hillel Yaffe Medical Center, Hadera, Hadera
  - Wolfson Medical Center, Holon
  - The Chaim Sheba Medical Center Tel Hashomer, Tel Hashomer, Ramat Gan
  - Sourasky Medical Center, Telaviv
- Italy (23):
  - Osp. SS Filippo Nicola, Avezzano
  - Policlinico S. Orsola Malpighi, Bologna
  - A.O. Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliero Universitaria di Ferrara, Cona (FE)
  - Policlinico San Martino, Genova
  - A.O.U.Policlinico G.Martino, Messina
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - Istituto Auxologico Italiano, Milan
  - Nuovo Ospedale Civile S. Agostino-Estense, Modena
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Ospedale S.Maria della Misericordia, AO di Perugia, Perugia
  - Osp. Guglielmo da Saliceto AUSL di Piacenza, Piacenza
  - Ospedale Santa Corona Azienda Sanitaria Locale n.2 Savonese, Pietra Ligure
  - Università degli Studi Campus Bio-Medico, Roma
  - A.O. San Camillo Forlanini, Roma
  - Umberto I Pol. di Roma-Università di Roma La Sapienza, Roma
  - Azienda Ospedaliera Sant'Andrea-Università di Roma La Sapienza, Roma
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
  - Ospedale Molinette, AO Città della Salute e della, Torino
  - Ospedale Maria Vittoria, Torino
  - Ospedale S. Maria di Ca' Foncello Azienda ULSS9 TREVISO, Treviso
  - A. O. Ospedale Circolo Fond. Macchi, Varese
  - Ospedale Policlinico G.B. Rossi (Borgo Roma) di Verona, Verona
- Japan (63):
  - Chubu Rosai Hospital, Aichi, Nagoya
  - National Hospital Organization Toyohashi Medical Center, Aichi, Toyohashi
  - Toyota Memorial Hospital, Aichi, Toyota
  - Reserch Institute for Brain and Blood Vessels Akita, Akita, Akita
  - Juntendo University Urayasu Hospital, Chiba, Urayasu
  - Go Neurosurgical Clinic, Fukuoka, Chikushi-gun
  - Fukuoka University Chikushi Hospital, Fukuoka, Chikushino
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Fukuoka Wajiro Hospital, Fukuoka, Fukuoka
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Fukuoka Tokushukai Medical Center, Fukuoka, Kasuga
  - Steel Memorial Yawata Hospital, Fukuoka, Kitakyushu
  - Japan Community Health Care Organization Kyushu Hospital, Fukuoka, Kitakyushu
  - St. Mary's Hospital, Fukuoka, Kurume
  - Shin Koga Hospital, Fukuoka, Kurume
  - Fukuoka Shin Mizumaki Hospital, Fukuoka, Onga
  - Social Insurance Tagawa Hospital, Fukuoka, Tagawa
  - Shin Yukuhashi Hospital, Fukuoka, Yukuhashi
  - Fujita General Hospital, Fukushima, Date-Gun
  - Shinseikai Masu Memorial Hospital, Fukushima, Nihonmatsu
  - Asahi University Hospital, Gifu, Gifu
  - Japanese Red Cross Takayama Hospital, Gifu, Takayama
  - Mihara Memorial Hospital, Gunma, Isesaki
  - Maebashi Red Cross Hospital, Gunma, Maebashi
  - Medical corporation Suiseikai Suiseikai Kajikawa Hospital, Hiroshima, Hiroshima
  - Araki Neurosurgical Hospital, Hiroshima, Hiroshima
  - Hiroshima Prefectural Hospital, Hiroshima, Hiroshima
  - Sapporo Shiroishi Memorial Hospital, Hokkaido, Sapporo
  - Nakamura Memorial Hospital, Hokkaido, Sapporo
  - Kobe City Medical Center General Hospital, Hyogo, Kobe
  - JA Toride Medical Center, Ibaraki, Toride
  - Tsukuba Medical Center Hospital, Ibaraki, Tsukuba
  - Iwate Medical University Hospital, Iwate, Morioka
  - Kagoshima City Hospital, Kagoshima, Kagoshima
  - National Hospital Organization Kagoshima Medical Center, Kagoshima, Kagoshima
  - Shonan Kamakura General Hospital, Kanagawa, Kamakura
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Japanese Red Cross Kumamoto Hospital, Kumamoto, Kumamoto
  - Kumamoto City Hospital, Kumamoto, Kumamoto
  - Uji-Tokushukai Medical Center, Kyoto, Uji
  - National Hospital Organization Sendai Medical Center, Miyagi, Sendai
  - South Miyagi Medical Center, Miyagi, Shibata-gun
  - Ina Central Hospital, Nagano, Ina
  - Nagano Municipal Hospital, Nagano, Naganoi
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Nozaki Tokushukai Hospital, Osaka, Daito
  - Higashiosaka City Medical Center, Osaka, Higashiosaka
  - Wakakusa Daiichi Hospital, Osaka, Higashiosaka
  - Rinku General Medical Center, Osaka, Izumisano
  - Kishiwada Tokushukai Hospital, Osaka, Kishiwada
  - Yagi Neurosurgical Hospital, Osaka, Osaka
  - Tominaga Hospital, Osaka, Osaka
  - Osaka University Hospital, Osaka, Suita
  - TMG Asaka Medical Center, Saitama, Asaka
  - Saitama Medical University International Medical Center, Saitama, Hidaka
  - Sainokuni Higashiomiya Medical Center, Saitama, Saitama
  - Saitama Municipal Hospital, Saitama, Saitama
  - Nippon Medical School Hospital, Tokyo, Bunkyo-ku
  - Tokyo Metropolitan Geriatric Hospital, Tokyo, Itabashi-ku
  - Kyorin University Hospital, Tokyo, Mitaka
  - Tokyo Women's Medical University Hospital, Tokyo, Shinjuku-ku
  - Saiseikai Wakayama Hospital, Wakayama, Wakayama
  - Yamagata City Hospital SAISEIKAN, Yamagata, Yamagata
- Malaysia (3):
  - Sarawak General Hospital, Kuching
  - Hospital Seberang Jaya, Pulau Pinang
  - Hospital Sultanah Nur Zahirah, Terengganu
- Mexico (5):
  - Hospital General de Culiacán "Dr. Bernardo J. Gastellum", Culiacán
  - Hospital Angeles del Pedregal, México, D.F.
  - Hospital General "Dr. Miguel Silva", Morelia
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Nuevo León
  - H. Central Dr Ignacio M. P., San Luis Potosí City
- New Zealand (3):
  - Auckland City Hospital, Grafton / Auckland
  - North Shore Hospital, Takapuna, Takpuna Auckland
  - Wellington Hospital, Wellington
- Peru (2):
  - Instituto Nacional de Ciencias Neurológicas, Barrios Altos
  - Hospital Nacional Guillermo Almenara Irigoyen, La Victoria
- Poland (10):
  - PI HOUSE Sp. z o.o., Gdansk, Gdansk
  - Spec.Hosp.of Dr. Wladyslaw Bieganski in Grudziadz, Grudziądz
  - Univ.Clin.Centr Gibinski of Silesian Med,Neurol.dep,Katowice, Katowice
  - University Hospital in Krakow, Krakow
  - Center of Clinical Neurology, private prac, Krakow, Krakow
  - Clin.Research Center,Leszek Szczepanski,Private Prac.,Lublin, Lublin
  - Medicome Sp. z o.o., Oświęcim
  - Specialist Holy Spirit Hospital, Neurology Dept,Sandomierz, Sandomierz
  - Public Central Clinical Hosp,Neurology Clinic,Warsaw, Warsaw
  - Military Institute of Medicine Neurology Clinic, Warsaw, Warsaw
- Portugal (12):
  - Hospital Garcia de Orta, EPE, Almada
  - Hospital Fernando Fonseca, EPE, Amadora
  - Hospital de Braga - Centro Clínico Académico (2CA), Braga
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - CHLC, EPE - Hospital de São José, Lisbon
  - CHLO, EPE - Hospital Egas Moniz, Lisbon
  - CHULN, EPE - Hospital de Santa Maria, Lisbon
  - Hospital Beatriz Ângelo, Loures
  - USLM, EPE - Hospital Pedro Hispano, Matosinhos Municipality
  - H. Santo António - Centro Hospitalar do Porto, Porto
  - Centro Hospitalar São João,EPE, Porto
  - Centro Hospitalar de Entre o Douro e Vouga, E.P.E. - Hospital de São Sebastião, Santa Maria da Feira
- Russia (13):
  - Interreg. Clinical & Diagnostic Center, Neurol. Dept., Kazan, Kazan'
  - Reg.Clin.Hosp#1 na S.V.Ochapovskiy,Neurology#1 Dep,Krasnodar, Krasnodar
  - City Clin.Emergency Hosp of Kursk, Neurology Department No.2, Kursk
  - Clin.Hosp#2,na.Semashko,Russ.Railways,Restorative Med&Rehab., Moscow
  - CityClin.Hosp na I.V.Davydovsky of Dept of Healthcare Moscow, Moscow
  - Research&Clini Cent Neuropsychiatry Dep. Healthcare,Moscow, Moscow
  - City Clin.Hosp#1na N.I.Pirogov,Dept of Healthcare of Moscow, Moscow
  - Ltd liabilityCom.CityNeurologic Cntr Sibneiromed,Novosibirsk, Novosibirsk
  - Research Inst. of Emerg. Med., Vascul. Center,St. Petersburg, Saint Petersburg
  - Military Medical Academy n.a. C. M. Kirov, St. Petersburg, Saint Petersburg
  - Saratov State Med.Univ na V.I.Razumovsky,FacultyTherapy Clin, Saratov
  - Reg.State Instit.of Healthc.Smolensk Reg.Clin.Hosp,Neurology, Smolensk
  - Sverdlovsk Reg.Clin.Hosp.No.1, Yekaterinburg
- Serbia (4):
  - Clinical Center of Serbia, Belgrade
  - Special Hosp.for Cerebrovascul.Disease,'Sveti Sava,Belgrade, Belgrade
  - Clinical Centre Nis, Niš
  - Clinical Center of Vojvodina, Novi Sad
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - National Neuroscience Institute, Singapore
- Slovakia (2):
  - Faculty Hospital L. Pasteura, Kosice, Košice
  - Faculty Hospital Nitra, Nitra
- Slovenia (3):
  - Instit.f.applicative Research in med.rehab.Dobrna, Dobrna
  - Cardial d.o.o., Specialist out-patient unit, Ljubljana, Ljubljana
  - Univ. Medical Center Maribor, Maribor
- South Africa (2):
  - University of Pretoria, Pretoria
  - Dr. Moodley and Dr. Sarvan, Tongaat
- South Korea (17):
  - Hallym University Sacred Heart Hospital, Anyang
  - Dong-A University Hospital, Busan
  - Kyungpook National Univ. Hosp, Daegu
  - Chungnam National University Hospital, Daejoen
  - Inje University Ilsan Paik Hospital, Goyang
  - Chonnam National University Hospital, Gwangju
  - Chosun University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Seongnam
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Samsung Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Ajou University Hospital, Suwon
- Spain (20):
  - Hospital General Universitario de Albacete, Albacete
  - Hospital del Mar, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Arnau de Vilanova, Lleida
  - Hospital La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital La Paz, Madrid
  - Hospital Son Espases, Palma de Mallorca
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Clínico de Santiago, Santiago de Compostela
  - Hospital Virgen del Rocío, Seville
  - Hospital Universitari Joan XXIII, Tarragona
  - Hospital Mútua Terrassa, Tarrasa (Barcelona)
  - Hospital Clínico de Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
- Sweden (5):
  - Sahlgrenska US, Göteborg, Gothenburg
  - Sahlgrenska Universitetssjukhuset, Östra, Gothenburg
  - Skaraborgs Sjukhus, Skövde
  - Karolinska Univ. sjukhuset, Stockholm
  - Danderyds Sjukhus, Stockholm
- Switzerland (7):
  - Canton Hospital Aarau, Neurology Dept., Stroke Center, Aarau
  - University Hospital Basel, Basel
  - Univ. Hospital Bern, Neurology Dept, Stroke Center, Bern
  - CHUV - Centre hospitalier universitaire vaudois, Lausanne
  - Regional Hospital Lugano,Neurocenter of Southern Switzerland, Lugano
  - Kantonsspital St.Gallen, Sankt Gallen
  - University Hosp. Zürich, Dept. of Neurology, Stroke Center, Zurich
- Taiwan (13):
  - Chang-Hua Christian Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - NCKUH, Tainan
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Cheng Hsin General Hospital, Taipei
  - Taipe Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital(TaoYuan), Taoyuan District
- Thailand (4):
  - Chulalongkorn University, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Lampang Hospital, Lampang
- Turkey (Türkiye) (14):
  - Ankara Universitesi Tip Fakultesi, Ankara
  - Hacettepe Universitesi Tip Fakultesi Noroloji A.B.D., Ankara
  - Gazi Universitesi Tip Fakultesi, Ankara
  - Eskisehir Osmangazi Universitesi Tip Fakultesi, Eskişehir
  - Bezmialem Vakif Universitesi Tip Fakultesi Hastanesi, Istanbul
  - Istanbul Universitesi Istanbul Tip Fakultesi Noroloji A.B.D., Istanbul
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Bakirkoy Prof. Dr. Mazhar Osman Ruh Sagligi ve Sinir Hastaliklari, Istanbul
  - Bakırkoy Dr. Sadi Konuk Egitim Ve Arastirma Hastanesi, Istanbul
  - Sisli Hamidiye Etfal Egitim ve Arastirma Hastanesi, Istanbul
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi, Istanbul
  - Dokuz Eylul Universitesi Tip Fakultesi Noroloji A.B.D., Izmir
  - Ondokuz Mayis Universitesi Tip Fakultesi, Samsun
  - Namik Kemal Universitesi Tip Fakultesi, Tekirdağ
- Ukraine (8):
  - Bukovinian Med.Univ.Chernivtsi Reg.Psychiatric Hosp,Neurolog, Chernivtsi
  - City Clinical Hospital No. 7, Kharkov, Kharkiv
  - Instit.of Neurol,Psychiatry&Narcol,Vascul. Malformations Dep, Kharkiv
  - Instit.of Gerontology na D.F.Chebotarev,Brain Vascular Path., Kyiv
  - Lviv Regional Clinical Hospital, Lviv, Lviv
  - Ternopil State Med.Univ.na Gorbachevskiy,Neurology Dept N3, Ternopil
  - Vinnitsia Reg.Psychoneurol.Hosp.na Yushchenko,Dept.N3,Neurol, Vinnitsia
  - Zhytomyr Reg.ClinHosp na Gerbachevskiy RegCouncil,Neurol.Dep, Zhytomyr

REFERENCES:
- [Derived] Del Brutto VJ, Diener HC, Easton JD, Granger CB, Cronin L, Kleine E, Grauer C, Brueckmann M, Toyoda K, Schellinger PD, Lyrer P, Molina CA, Chutinet A, Bladin CF, Estol CJ, Sacco RL. Predictors of Recurrent Stroke After Embolic Stroke of Undetermined Source in the RE-SPECT ESUS Trial. J Am Heart Assoc. 2022 Jun 7;11(11):e023545. doi: 10.1161/JAHA.121.023545. Epub 2022 Jun 3. PMID 35656979
- [Derived] Diener HC, Easton JD, Hart RG, Kasner S, Kamel H, Ntaios G. Review and update of the concept of embolic stroke of undetermined source. Nat Rev Neurol. 2022 Aug;18(8):455-465. doi: 10.1038/s41582-022-00663-4. Epub 2022 May 10. PMID 35538232
- [Derived] Bahit MC, Sacco RL, Easton JD, Meyerhoff J, Cronin L, Kleine E, Grauer C, Brueckmann M, Diener HC, Lopes RD, Brainin M, Lyrer P, Wachter R, Segura T, Granger CB; RE-SPECT ESUS Steering Committee and Investigators. Predictors of Atrial Fibrillation Development in Patients With Embolic Stroke of Undetermined Source: An Analysis of the RE-SPECT ESUS Trial. Circulation. 2021 Nov 30;144(22):1738-1746. doi: 10.1161/CIRCULATIONAHA.121.055176. Epub 2021 Oct 15. PMID 34649459
- [Derived] Uchiyama S, Toyoda K, Lee BC, Liou CW, Wong LKS, Grauer C, Brueckmann M, Taniguchi A, Urano Y, Easton JD; RE-SPECT ESUS Investigators. Dabigatran or Aspirin in East Asian Patients With Embolic Stroke of Undetermined Source: RE-SPECT ESUS Subgroup Analysis. Stroke. 2021 Mar;52(3):1069-1073. doi: 10.1161/STROKEAHA.120.031891. Epub 2021 Feb 16. PMID 33588594
- [Derived] Diener HC, Chutinet A, Easton JD, Granger CB, Kleine E, Marquardt L, Meyerhoff J, Zini A, Sacco RL. Dabigatran or Aspirin After Embolic Stroke of Undetermined Source in Patients With Patent Foramen Ovale: Results From RE-SPECT ESUS. Stroke. 2021 Mar;52(3):1065-1068. doi: 10.1161/STROKEAHA.120.031237. Epub 2021 Jan 28. PMID 33504190
- [Derived] Diener HC, Sacco RL, Easton JD, Granger CB, Bar M, Bernstein RA, Brainin M, Brueckmann M, Cronin L, Donnan G, Gdovinova Z, Grauer C, Kleine E, Kleinig TJ, Lyrer P, Martins S, Meyerhoff J, Milling T, Pfeilschifter W, Poli S, Reif M, Rose DZ, Sanak D, Schabitz WR. Antithrombotic Treatment of Embolic Stroke of Undetermined Source: RE-SPECT ESUS Elderly and Renally Impaired Subgroups. Stroke. 2020 Jun;51(6):1758-1765. doi: 10.1161/STROKEAHA.119.028643. Epub 2020 May 14. PMID 32404035
- [Derived] Diener HC, Sacco RL, Easton JD, Granger CB, Bernstein RA, Uchiyama S, Kreuzer J, Cronin L, Cotton D, Grauer C, Brueckmann M, Chernyatina M, Donnan G, Ferro JM, Grond M, Kallmunzer B, Krupinski J, Lee BC, Lemmens R, Masjuan J, Odinak M, Saver JL, Schellinger PD, Toni D, Toyoda K; RE-SPECT ESUS Steering Committee and Investigators. Dabigatran for Prevention of Stroke after Embolic Stroke of Undetermined Source. N Engl J Med. 2019 May 16;380(20):1906-1917. doi: 10.1056/NEJMoa1813959. PMID 31091372

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was randomised, active comparator, double-blind, 2 arms (1:1 ratio) event-driven Phase III trial in participants with embolic stroke of undetermined source (ESUS). Study was conducted at multiple centers in 42 countries between 3 Dec 2014 (first participant enrollment) and 14 August 2018 (last participant visit).
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist sites which would then ensured that all participants met all inclusion/exclusion criteria. Participants were not to be randomized to trial treatment if any one of the specific entry criteria were not met.
Groups:
- Dabigatran Etexilate 110 or 150 Milligram (mg): Participants were orally administered one 110 mg (for participants aged ≥75 years or with a creatinine clearance (CrCl) of 30 to <50 millilitre/ minute (mL/min)) or one 150 mg (for participants aged <75 years and with a CrCl of ≥50 mL/minute) Dabigatran etexilate (DE) capsule twice daily.
- Acetylsalicylic Acid, Aspirin (ASA) 100 mg: Participants were orally administered one 100 mg Aspirin non-enteric coated tablet once daily.
Period: Overall Study
Arm/Group | Dabigatran Etexilate 110 or 150 Milligram (mg) | Acetylsalicylic Acid, Aspirin (ASA) 100 mg
Started (Randomised) | 2695 | 2695
Completed | 2620 | 2623
Not Completed | 75 | 72
Not completed — Death | 56 | 58
Not completed — Lost to Follow-up | 19 | 14

BASELINE CHARACTERISTICS:
Population: Randomised set (RS): The RS consisted of all patients who were randomised, regardless of whether they took trial medication. The start date of the observation period for this population was the date of randomisation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran Etexilate 110 or 150 Milligram (mg) | Acetylsalicylic Acid, Aspirin (ASA) 100 mg | Total
Number analyzed (Participants) | 2695 | 2695 | 5390
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (11.44) | 63.9 (11.39) | 64.2 (11.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1001 | 986 | 1987
  Male | 1694 | 1709 | 3403
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Information on race and ethnicity was not collected for all patients in France.
  Participants
    Hispanic or Latino | 281 | 268 | 549
    Not Hispanic or Latino | 2354 | 2371 | 4725
    Unknown or Not Reported | 60 | 56 | 116
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 20 | 31
  Asian | 631 | 597 | 1228
  Native Hawaiian or Other Pacific Islander | 2 | 4 | 6
  Black or African American | 54 | 40 | 94
  White | 1926 | 1966 | 3892
  More than one race | 10 | 12 | 22
  Unknown or Not Reported | 61 | 56 | 117

OUTCOME MEASURES:

1. Primary Outcome: Adjudicated Recurrent Stroke
Description: Adjudicated recurrent stroke (ischemic, hemorrhagic, or unspecified) is presented. The annualised event rate represents the average number of events per patient during a 1-year period.
Time Frame: From randomisation until full follow up period, approximately 43 months.
Population: Randomised set (RS): RS consisted of all participants who were randomised, regardless of whether they took trial medication. The start date of the observation period for this population was the date of randomisation.
Measure: Number; unit: Annualised event rate (%/ year)
Arm/Group | Dabigatran Etexilate 110 or 150 Milligram (mg) | Acetylsalicylic Acid, Aspirin (ASA) 100 mg
Number analyzed (Participants) | 2695 | 2695
Annualised event rate (%/ year) | 4.09 | 4.80
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110 or 150 Milligram (mg) vs Acetylsalicylic Acid, Aspirin (ASA) 100 mg; Test type: Superiority; p = 0.1028, Regression, Cox; Covariates in model are age(<or>= 75years), creatinine clearance < or >= 50mL/min and stroke or transient ischaemic attack(TIA) prior to index stroke; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.69 to 1.03]

2. Primary Outcome: First Major Bleed (Adjudicated)
Description: First major bleed is primary safety endpoint. Major bleeds were defined according to the International Society of Thrombosis and Haemostasis (ISTH) definition as follows:
  * Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome and/or,
  * Bleeding (which should be overt) associated with a reduction in haemoglobin of at least 2 grams/ decilitre (g/dL) (1.24 millimoles Per Litre (mmol/L)), or leading to transfusion of ≥2 units of blood or packed cells (equivalent to ≥4.5 units in Japan); the haemoglobin drop should be considered to be due to and temporally related to the bleeding event and/or,
  * Fatal bleed. The annualised event rate represents the average number of events per patient during a 1-year period.
Time Frame: Between the first trial medication intake up to 6 days after the last trial medication intake, approximately 42 months.
Population: Treated set (TS): TS consisted of all patients who were treated with at least 1 dose of trial medication. The start date of the observation period for this population was the date of first intake of trial medication.
Measure: Number; unit: Annualised event rate (%/ year)
Arm/Group | Dabigatran Etexilate 110 or 150 Milligram (mg) | Acetylsalicylic Acid, Aspirin (ASA) 100 mg
Number analyzed (Participants) | 2676 | 2674
Annualised event rate (%/ year) | 1.84 | 1.33
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110 or 150 Milligram (mg) vs Acetylsalicylic Acid, Aspirin (ASA) 100 mg; Test type: Superiority; p = 0.1076, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.36, 95% CI 2-sided [0.94 to 1.97]

3. Secondary Outcome: Adjudicated Ischaemic Stroke
Description: Adjudicated ischaemic stroke is a key secondary endpoint. The annualised event rate represents the average number of events per patient during a 1-year period.
Time Frame: From randomisation until full follow up period, up to 43 months
Population: RS
Measure: Number; unit: Annualised event rate (%/ year)
Arm/Group | Dabigatran Etexilate 110 or 150 Milligram (mg) | Acetylsalicylic Acid, Aspirin (ASA) 100 mg
Number analyzed (Participants) | 2695 | 2695
Annualised event rate (%/ year) | 3.97 | 4.71
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110 or 150 Milligram (mg) vs Acetylsalicylic Acid, Aspirin (ASA) 100 mg; Test type: Superiority; p = 0.0892, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.68 to 1.03]

4. Secondary Outcome: Adjudicated Composite of Non-fatal Stroke, Non-fatal Myocardial Infarction, or Cardiovascular Death
Description: Adjudicated composite of non-fatal stroke, non-fatal myocardial infarction (MI), or cardiovascular death is a key secondary endpoint. The annualised event rate represents the average number of events per patient during a 1-year period.
Time Frame: From randomisation until full follow up period, up to 43 months
Population: RS
Measure: Number; unit: Annualised event rate (%/ year)
Arm/Group | Dabigatran Etexilate 110 or 150 Milligram (mg) | Acetylsalicylic Acid, Aspirin (ASA) 100 mg
Number analyzed (Participants) | 2695 | 2695
Annualised event rate (%/ year) | 4.80 | 5.40
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110 or 150 Milligram (mg) vs Acetylsalicylic Acid, Aspirin (ASA) 100 mg; Test type: Superiority; p = 0.1911, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.73 to 1.06]

5. Secondary Outcome: Disabling Stroke
Description: Disabling stroke (modified Rankin Scale greater than or equal to 4, as determined 3 months after recurrent stroke) is presented. The annualised event rate represents the average number of events per patient during a 1-year period.
Time Frame: From randomisation until full follow up period, up to 43 months
Population: RS
Measure: Number; unit: Annualised event rate (%/ year)
Arm/Group | Dabigatran Etexilate 110 or 150 Milligram (mg) | Acetylsalicylic Acid, Aspirin (ASA) 100 mg
Number analyzed (Participants) | 2695 | 2695
Annualised event rate (%/ year) | 0.55 | 0.93
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110 or 150 Milligram (mg) vs Acetylsalicylic Acid, Aspirin (ASA) 100 mg; Test type: Superiority; p = 0.0354, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.36 to 0.96]

6. Secondary Outcome: All-cause Death
Description: All-cause death is presented. The annualised event rate represents the average number of events per patient during a 1-year period.
Time Frame: From randomisation until full follow up period, up to 43 months
Population: RS
Measure: Number; unit: Annualised event rate (%/ year)
Arm/Group | Dabigatran Etexilate 110 or 150 Milligram (mg) | Acetylsalicylic Acid, Aspirin (ASA) 100 mg
Number analyzed (Participants) | 2695 | 2695
Annualised event rate (%/ year) | 1.24 | 1.28
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110 or 150 Milligram (mg) vs Acetylsalicylic Acid, Aspirin (ASA) 100 mg; Test type: Superiority; p = 0.8074, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.66 to 1.38]

7. Secondary Outcome: Adjudicated Intracranial Hemorrhage
Description: Adjudicated intracranial haemorrhage comprised the subtypes of intracerebral bleeds, intraventricular bleeds, subdural bleeds, epidural bleeds, and subarachnoid bleeds. Microbleeds did not qualify as intracranial haemorrhage, except when they were symptomatic.
  The annualised event rate represents the average number of events per patient during a 1-year period.
Time Frame: Between the first trial medication intake up to 6 days after the last trial medication intake, approximately 42 months.
Population: TS
Measure: Number; unit: Annualised event rate (%/ year)
Arm/Group | Dabigatran Etexilate 110 or 150 Milligram (mg) | Acetylsalicylic Acid, Aspirin (ASA) 100 mg
Number analyzed (Participants) | 2676 | 2674
Annualised event rate (%/ year) | 0.67 | 0.63
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110 or 150 Milligram (mg) vs Acetylsalicylic Acid, Aspirin (ASA) 100 mg; Test type: Superiority; p = 0.9064, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.58 to 1.83]

8. Secondary Outcome: Adjudicated Fatal Bleed
Description: Adjudicated fatal bleeding was defined as a bleeding event which the Independent Event Adjudication Committee (IAC) determined as the primary cause of death or contributed directly to death. The annualised event rate represents the average number of events per patient during a 1-year period. Because there were 0 events in one treatment group, the hazard ratio is unable to be calculated.
Time Frame: Between the first trial medication intake up to 6 days after the last trial medication intake, approximately 42 months.
Population: TS
Measure: Number; unit: Annualised event rate (%/ year)
Arm/Group | Dabigatran Etexilate 110 or 150 Milligram (mg) | Acetylsalicylic Acid, Aspirin (ASA) 100 mg
Number analyzed (Participants) | 2676 | 2674
Annualised event rate (%/ year) | 0.00 | 0.05

9. Secondary Outcome: Adjudicated Life-threatening Bleed
Description: Major bleeds were to be classified as life-threatening if they met one or more of the following criteria: fatal bleed, symptomatic intracranial bleed, reduction in haemoglobin of at least 5 grams/ deciliter (g/dL), transfusion of at least 4 units of packed red blood cells (equivalent to 9 units in Japan), associated with hypotension requiring the use of intravenous inotropic agents, or necessitated surgical intervention.
  The annualised event rate represents the average number of events per patient during a 1-year period.
Time Frame: Between the first trial medication intake up to 6 days after the last trial medication intake, approximately 42 months.
Population: TS
Measure: Number; unit: Annualised event rate (%/ year)
Arm/Group | Dabigatran Etexilate 110 or 150 Milligram (mg) | Acetylsalicylic Acid, Aspirin (ASA) 100 mg
Number analyzed (Participants) | 2676 | 2674
Annualised event rate (%/ year) | 0.76 | 0.91
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110 or 150 Milligram (mg) vs Acetylsalicylic Acid, Aspirin (ASA) 100 mg; Test type: Superiority; p = 0.4352, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.49 to 1.36]

10. Secondary Outcome: Any Bleed (Investigator-reported)
Description: This was the sum of all major and minor bleeds (Minor bleeds were clinical bleeds that did not fulfil the criteria for major bleeds), regardless of severity.
  The annualised event rate represents the average number of events per patient during a 1-year period.
Time Frame: Between the first trial medication intake up to 6 days after the last trial medication intake, approximately 42 months.
Population: TS
Measure: Number; unit: Annualised event rate (%/ year)
Arm/Group | Dabigatran Etexilate 110 or 150 Milligram (mg) | Acetylsalicylic Acid, Aspirin (ASA) 100 mg
Number analyzed (Participants) | 2676 | 2674
Annualised event rate (%/ year) | 15.21 | 11.64
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110 or 150 Milligram (mg) vs Acetylsalicylic Acid, Aspirin (ASA) 100 mg; Test type: Superiority; p = 0.0003, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.28, 95% CI 2-sided [1.12 to 1.47]

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) and serious AE starting between the first trial medication intake up to 6 days after the last trial medication intake, approximately 42 months. All-cause mortality reported from randomisation until full follow up period, approximately 43 months.
Description: All-cause mortality numbers are based on randomized set whereas Serious Adverse Events (SAE) and non-SAE are based on treated set.
Arm/Group | Dabigatran Etexilate 110 or 150 Milligram (mg) | Acetylsalicylic Acid, Aspirin (ASA) 100 mg
All-Cause Mortality (participants affected / at risk) | 56/2695 | 58/2695
Serious Adverse Events (participants affected / at risk) | 724/2676 | 740/2674
Other Adverse Events (participants affected / at risk) | 306/2676 | 295/2674
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate 110 or 150 Milligram (mg) (N=2676) | Acetylsalicylic Acid, Aspirin (ASA) 100 mg (N=2674)
Anaemia (Blood and lymphatic system disorders) | 7 | 3
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 11 | 8
Angina pectoris (Cardiac disorders) | 3 | 4
Angina unstable (Cardiac disorders) | 4 | 2
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 24 | 20
Atrial fibrillation or atrial flutter (Cardiac disorders) | 34 | 29
Atrial flutter (Cardiac disorders) | 10 | 10
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 5 | 10
Cardiac failure acute (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 4 | 2
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 6 | 11
Coronary artery stenosis (Cardiac disorders) | 0 | 3
Myocardial infarction (Cardiac disorders) | 8 | 8
Prinzmetal angina (Cardiac disorders) | 2 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Heart disease congenital (Congenital, familial and genetic disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 2 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 2 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 6 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 4 | 7
Diabetic retinopathy (Eye disorders) | 1 | 0
Eye haemorrhage (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 6 | 6
Macular degeneration (Eye disorders) | 3 | 2
Macular fibrosis (Eye disorders) | 1 | 2
Pterygium (Eye disorders) | 0 | 1
Retinal drusen (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Colitis (Gastrointestinal disorders) | 0 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 2 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 5 | 3
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ischaemic enteritis (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 2 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Rectal perforation (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3
Bile duct stone (Hepatobiliary disorders) | 0 | 3
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 3 | 1
Cholelithiasis (Hepatobiliary disorders) | 4 | 3
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 2
Bronchitis (Infections and infestations) | 2 | 1
Bronchitis bacterial (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 3 | 1
Erysipelas (Infections and infestations) | 2 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 5 | 4
Periodontitis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 2 | 2
Pneumonia (Infections and infestations) | 18 | 14
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 3 | 4
Sepsis (Infections and infestations) | 5 | 6
Tuberculous pleurisy (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 13 | 5
Airway burns (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 4 | 2
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 21 | 9
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 1
Femur fracture (Injury, poisoning and procedural complications) | 3 | 2
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 2
Meniscus injury (Injury, poisoning and procedural complications) | 4 | 2
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 1
Near drowning (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 4
Rib fracture (Injury, poisoning and procedural complications) | 4 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 3
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 2 | 4
Subdural haematoma (Injury, poisoning and procedural complications) | 7 | 3
Subdural haemorrhage (Injury, poisoning and procedural complications) | 3 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 3
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Creatinine renal clearance decreased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Diffuse idiopathic skeletal hyperostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 4
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 | 19
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 12
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebellar haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 2
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 6
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain stem infarction (Nervous system disorders) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 3
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 25 | 42
Cerebrovascular accident (Nervous system disorders) | 95 | 97
Diplegia (Nervous system disorders) | 0 | 1
Embolic cerebral infarction (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 1 | 2
Epilepsy (Nervous system disorders) | 18 | 25
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 3
Hemianaesthesia (Nervous system disorders) | 2 | 2
Hemiparesis (Nervous system disorders) | 5 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 4
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 2
Ischaemic stroke (Nervous system disorders) | 47 | 45
Lacunar infarction (Nervous system disorders) | 0 | 1
Multiple sclerosis (Nervous system disorders) | 1 | 0
Muscle spasticity (Nervous system disorders) | 0 | 1
Post stroke seizure (Nervous system disorders) | 3 | 0
Seizure (Nervous system disorders) | 17 | 16
Temporal lobe epilepsy (Nervous system disorders) | 0 | 1
Thrombotic cerebral infarction (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 46 | 41
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 2
Adjustment disorder (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 2
Bipolar disorder (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 5 | 2
Depression (Psychiatric disorders) | 7 | 4
Major depression (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 3
Acute kidney injury (Renal and urinary disorders) | 8 | 10
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 6 | 5
Pollakiuria (Renal and urinary disorders) | 0 | 1
Postrenal failure (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 4
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 5 | 3
Prostatitis (Reproductive system and breast disorders) | 2 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 4 | 9
Ischaemia (Vascular disorders) | 0 | 3
Peripheral artery occlusion (Vascular disorders) | 1 | 5
Asthenia (General disorders) | 2 | 1
Chest pain (General disorders) | 7 | 5
Pyrexia (General disorders) | 2 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 2
Atrial tachycardia (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 2 | 1
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 3 | 5
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 2 | 0
Palpitations (Cardiac disorders) | 2 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1
Sinoatrial block (Cardiac disorders) | 1 | 0
Sinus arrest (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 3
Atrial septal defect (Congenital, familial and genetic disorders) | 3 | 4
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 | 1
Cryopyrin associated periodic syndrome (Congenital, familial and genetic disorders) | 1 | 0
Factor V Leiden mutation (Congenital, familial and genetic disorders) | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 4 | 1
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 7 | 8
Vertigo positional (Ear and labyrinth disorders) | 3 | 3
Adrenal haematoma (Endocrine disorders) | 1 | 0
Adrenal mass (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Toxic nodular goitre (Endocrine disorders) | 1 | 0
Age-related macular degeneration (Eye disorders) | 1 | 0
Amaurosis (Eye disorders) | 0 | 1
Amaurosis fugax (Eye disorders) | 3 | 1
Angle closure glaucoma (Eye disorders) | 0 | 1
Blepharitis (Eye disorders) | 1 | 0
Cataract nuclear (Eye disorders) | 1 | 0
Dacryostenosis acquired (Eye disorders) | 1 | 0
Idiopathic orbital inflammation (Eye disorders) | 1 | 0
Macular hole (Eye disorders) | 0 | 1
Narrow anterior chamber angle (Eye disorders) | 0 | 1
Optic atrophy (Eye disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 2 | 0
Retinal detachment (Eye disorders) | 0 | 1
Retinal tear (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Appendix disorder (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 | 5
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileal perforation (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 3
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intestinal polyp (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Subileus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest discomfort (General disorders) | 1 | 0
Death (General disorders) | 3 | 6
Fatigue (General disorders) | 1 | 1
Feeling cold (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 2
General physical health deterioration (General disorders) | 1 | 0
Ill-defined disorder (General disorders) | 1 | 0
Incarcerated hernia (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 3
Necrosis (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 0
Sudden cardiac death (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Vascular stent stenosis (General disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Appendiceal abscess (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 2
Conjunctivitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 2 | 0
Ear infection (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 2
Epididymitis (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 3 | 2
Gastroenteritis norovirus (Infections and infestations) | 1 | 1
Haematoma infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 0
Leptospirosis (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 1 | 0
Mycotoxicosis (Infections and infestations) | 0 | 1
Neuroborreliosis (Infections and infestations) | 1 | 0
Neurosyphilis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 2
Otitis media acute (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 0 | 1
Perineal abscess (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1
Pulpitis dental (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 2 | 3
Septic embolus (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 2 | 0
Sialoadenitis (Infections and infestations) | 1 | 0
Thrombophlebitis septic (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 1 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 2 | 2
Exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2
Injury (Injury, poisoning and procedural complications) | 2 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 3
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Poisoning deliberate (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 1
Bile duct pressure increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Computerised tomogram thorax abnormal (Investigations) | 0 | 1
Electrocardiogram Q waves (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Influenza A virus test positive (Investigations) | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Necrotising myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Systemic scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian epithelial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour obstruction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aphasia (Nervous system disorders) | 2 | 2
Ataxia (Nervous system disorders) | 1 | 0
Brain injury (Nervous system disorders) | 1 | 0
Brain stem stroke (Nervous system disorders) | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0
Carotid artery aneurysm (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 3 | 3
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Central pain syndrome (Nervous system disorders) | 1 | 0
Cerebellar stroke (Nervous system disorders) | 1 | 0
Cerebral cyst (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 1
Cerebral vasoconstriction (Nervous system disorders) | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Cervicogenic headache (Nervous system disorders) | 0 | 1
Cubital tunnel syndrome (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 1 | 2
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 8 | 4
Dizziness postural (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 2 | 1
Facial paralysis (Nervous system disorders) | 0 | 3
Facial paresis (Nervous system disorders) | 0 | 1
Focal dyscognitive seizures (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 2 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Haemorrhagic transformation stroke (Nervous system disorders) | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 2 | 2
Migraine with aura (Nervous system disorders) | 1 | 1
Monoparesis (Nervous system disorders) | 1 | 0
Monoplegia (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 1
Neuralgic amyotrophy (Nervous system disorders) | 1 | 0
Neurodegenerative disorder (Nervous system disorders) | 0 | 1
Neuroglycopenia (Nervous system disorders) | 1 | 0
Neurological symptom (Nervous system disorders) | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 2 | 2
Partial seizures (Nervous system disorders) | 5 | 5
Polyneuropathy (Nervous system disorders) | 0 | 1
Post stroke epilepsy (Nervous system disorders) | 2 | 2
Presyncope (Nervous system disorders) | 1 | 0
Pseudostroke (Nervous system disorders) | 0 | 1
Radial nerve compression (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 2 | 2
Sensory disturbance (Nervous system disorders) | 0 | 1
Sensory loss (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 3 | 1
Syncope (Nervous system disorders) | 8 | 6
Tonic convulsion (Nervous system disorders) | 0 | 1
Transient global amnesia (Nervous system disorders) | 0 | 2
Visual field defect (Nervous system disorders) | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 2
Device dislocation (Product Issues) | 0 | 1
Aggression (Psychiatric disorders) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 1
Generalised anxiety disorder (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 1
Post stroke depression (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Somatic symptom disorder (Psychiatric disorders) | 0 | 1
Anuria (Renal and urinary disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 3 | 0
Calculus urinary (Renal and urinary disorders) | 3 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Glomerulonephritis proliferative (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 6 | 3
Renal colic (Renal and urinary disorders) | 1 | 3
Renal failure (Renal and urinary disorders) | 4 | 1
Renal impairment (Renal and urinary disorders) | 0 | 2
Renal ischaemia (Renal and urinary disorders) | 0 | 1
Renal mass (Renal and urinary disorders) | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Urogenital haemorrhage (Renal and urinary disorders) | 1 | 0
Acquired hydrocele (Reproductive system and breast disorders) | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Cervical polyp (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 3 | 0
Spermatocele (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Vaginal polyp (Reproductive system and breast disorders) | 1 | 0
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 2 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Tanning (Social circumstances) | 1 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 1
Hysterectomy (Surgical and medical procedures) | 0 | 1
Myomectomy (Surgical and medical procedures) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 2
Aortic occlusion (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Arteritis (Vascular disorders) | 1 | 0
Blue toe syndrome (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 2 | 1
Embolism (Vascular disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 0
Hypertensive crisis (Vascular disorders) | 11 | 4
Hypotension (Vascular disorders) | 0 | 2
Iliac artery occlusion (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 4
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 3
Shock haemorrhagic (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1
Vasospasm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate 110 or 150 Milligram (mg) (N=2676) | Acetylsalicylic Acid, Aspirin (ASA) 100 mg (N=2674)
Nasopharyngitis (Infections and infestations) | 173 | 170
Atrial fibrillation (Cardiac disorders) | 136 | 128

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT02239120/SAP_000.pdf
  • Study Protocol (2016-04-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT02239120/Prot_001.pdf